CLINICAL TRIAL: NCT05296603
Title: Efficacy and Biomarker Explanation of IBI-322 Plus Lenvatinib on Extensive Stage Small Cell Lung Cancer Who Failed From First Line PD-(L)-1 Inhibitors: Multiple Cohorts Perspective Study
Brief Title: Efficacy and Biomarker Explanation of IBI-322 Plus Lenvatinib on Extensive Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BELIEVE
Record Dates: First submitted 2022-03-15; First posted 2022-03-25 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Duration of response time less than 3 months
  Interventions: Drug: IBI-322 Plus Lenvatinib
- Cohort B (Experimental): Duration of response time between 3 and 6 months
  Interventions: Drug: IBI-322 Plus Lenvatinib
- Cohort C (Experimental): Duration of response time more than 6 months
  Interventions: Drug: IBI-322 Plus Lenvatinib

INTERVENTIONS:
Drug: IBI-322 Plus Lenvatinib — IBI322 is based on the "3+3" model, with a dose ascent starting from 10mg

SUMMARY:
This study aimed to explore the efficacy and biomarker explanation of IBI-322 Plus Lenvatinib on extensive stage small cell lung cancer who failed from first line PD-(L)1 inhibitors.

ELIGIBILITY:
* Eligible subjects selected for this study must meet all of the following criteria:

  1. Sign written informed consent before implementing any trial-related procedures;
  2. Age ≥18 years old and ≤75 years old;
  3. No limit on the gender;
  4. Patients with extensive stage SCLC diagnosed by pathology (as staged by the American Veterans Lung Cancer Association (VALG)), who do not have an imaging response during first-line treatment with PD-(L)1 inhibitors, or who progress after imaging reactions on first-line therapy (the most recent regimen prior to enrollment must contain PD-(L)1 inhibitors);
  5. According to the Response Evaluation Criteria for Solid Tumors (RECIST V1.1), there must be at least one lesion that can be measured by imaging. Lesions located within the radiation field of previous radiation therapy can be considered as measurable lesions if progress is confirmed;
  6. ECOG score 0-1 points;
  7. Expected survival time> 3 months;
  8. Sufficient organ function, subjects need to meet the following laboratory indicators:

  <!-- -->

  1. The absolute value of neutrophils (ANC) ≥1.5x109/L when no granulocyte colony-stimulating factor is used in the past 14 days;
  2. In the case of no blood transfusion in the past 14 days, platelets ≥100×109/L;
  3. In the past 14 days without blood transfusion or erythropoietin, hemoglobin>9g/dL;
  4. Total bilirubin≤1.5×upper limit of normal (ULN);
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) within ≤2.5×ULN (subjects with liver metastases are allowed to have ALT or AST ≤5×ULN);
  6. Serum creatinine ≤1.5×ULN and creatinine clearance rate (calculated by Cockcroft-Gault formula) ≥50ml/min;
  7. Good coagulation function, defined as International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times ULN;
  8. Normal thyroid function is defined as thyroid-stimulating hormone (TSH) within the normal range. If the baseline TSH is out of the normal range, subjects whose total T3 (or FT3) and FT4 are within the normal range can also be included in the group;
  9. Myocardial enzyme spectrum is within the normal range (for example, simple laboratory abnormalities that are judged by the investigator to be of no clinical significance are also allowed to be included in the group).

Exclusion Criteria:

* Patients with contraindication of chemotherapy Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
ORR | 12 weeks
  Defined as the proportion of subjects in complete remission (CR) and partial remission (PR) to the total subjects

SECONDARY OUTCOMES:
PFS | 1year
  Defined as the time from the beginning of treatment to the first imaging disease progression or death (whichever occurs first)
OS | 1 year
  Defined as the time from the start of treatment to the death of the subject due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China